CLINICAL TRIAL: NCT00695604
Title: Repeated High-dose Inhaled Corticosteroids for Asthma
Acronym: ReHICS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was not able to be completed, no results analyzed.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15322B
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Asthma
Keywords: Acute asthma; fluticasone; inhaled corticosteroids
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Placebo Comparator
  All patients assigned to this group will receive:
  1. Placebo via Metered Dose Inhaler (MDI).
  2. Albuterol via MDI.
  Interventions: Drug: Placebo
- 2 (Active Comparator): Active Comparator
  All patients assigned to this group will receive:
  1. Fluticasone via MDI.
  2. Albuterol via MDI.
  Interventions: Drug: Fluticasone

INTERVENTIONS:
Drug: Placebo — Placebo via MDI.
  Arms: 1
Drug: Fluticasone — Fluticasone MDI.
  Arms: 2

SUMMARY:
The purpose of this study is to to compare the effects of high-dose Inhaled Corticosteroids (ICS) vs. placebo in adults with chronic stable asthma.

ELIGIBILITY:
Inclusion criteria:

* Physician diagnosis of asthma.
* Age ≥18 years and ≤50 years
* Evidence of airflow obstruction as measured by spirometry and flow-volume loop per American Thoracic Society guidelines.
* Treatment for asthma with:

  * daily inhaled corticosteroids and long-acting beta2-agonists, AND
  * as-needed use of a short-acting beta2-agonist

Exclusion criteria:

* History of >10 pack-year tobacco use
* Other pulmonary or cardiac diagnosis that is actively being treated
* History of adverse events or allergy to fluticasone
* Systemic corticosteroid therapy within 7 days of study visit
* Inability to obtain written informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Airflow inflammation. | Pre-study and post-study drug administration

SECONDARY OUTCOMES:
Airflow obstruction. | Pre-study and post-study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Krishnan, MD, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States